CLINICAL TRIAL: NCT05569863
Title: Digital Pattern Recognition for Identification of Various Hypospadias Parameters Based on Digital Photography Using Artificial Neural Network
Brief Title: Identification of Hypospadias Parameters Using Digital Photography and Artificial Intelligence
Acronym: ASHOKA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Irfan Wahyudi, MD, PhD, Dr. dr. Irfan Wahyudi, Sp.U(K), Indonesia University
Other Study IDs: 22-03-0310; NKB-1235/UN2.RST/HKP.05.00 (Other Grant/Funding Number: Universitas Indonesia); KET-413/UN2.F1/ETIK/PPM.00.02 (Other: Faculty of Medicine, University of Indonesia)
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Hypospadias
Keywords: artificial intelligence; digital recognition; digital photography; hypospadias; machine learning
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypospadias group: Patients with hypospadias diagnosis
- Control group: Patients without hypospadias

SUMMARY:
The goal of this observational study is to develop and validate a digital pattern recognition system based on artificial neural network to determine various parameters in hypospadias. The main question it aims to answer is:

How accurate is the digital pattern recognition system based on artificial neural network to determine various parameters in hypospadias?

Participants in this study are hypospadias patients aged < 18 years old. The guardian (and the patient, if applicable) will be informed about the study and asked for consent. The digital picture of participants' penis will be taken from different angles according to the predetermined angle.

The clinical characteristics of the photographed penis are then inputted and used to train a customized artificial neural network (ANN). The machine is then used to predict various hypospadias parameters presenting at the patients' penis. The accuracy of the machine is then compared to the measurement done by pediatric urologists.

DETAILED DESCRIPTION:
This is a development protocol for a digital pattern recognition program for identification of various hypospadias parameters using artificial neural network. The population for this study are children suspected of having hypospadias who are admitted or referred to hospitals in Indonesia.

The consent for the capture of the images needed in the study will be obtained from the parents of hypospadias patients as part of the standard of care to be used as a clinical reference. The photograph taken for this study were kept in an encrypted database. The inclusion criteria of this study are children aged <18 years old who are suspected of having hypospadias, with age-matched control. Those with history of hypospadias repair or those who refuse to participate in the study are excluded.

The clinical outcomes measured in this study are:

1. Hypospadias status: hypospadias or non-hypospadias
2. Meatal location: glanular, coronal, distal shaft, proximal shaft, penoscrotal
3. Meatal shape: normal, abnormal
4. Quality of the urethral plate: good, bad
5. Glans diameter: in mm
6. Glans shape: normal, abnormal The clinical outcomes were measured preoperatively and 1 month postoperatively

A hypospadias and normal penis image with matched age database was used to train the artificial neural network. Three image aspects of the penis (ventral, dorsal, and lateral aspect which include the glans, shaft, and scrotum) were taken from each subjects. The data was labeled with hypospadias parameters: hypospadias status, meatal location, meatal shape, quality of the urethral plate, glans diameter, and glans shape. The data were uploaded to train the artificial neural network.

The statistical analysis plan will be followed for all clinical outcomes analyses. Standard error, 95% confidence intervals, and P values will be reported whenever possible. Intra and inter rater analysis will be performed using the Fleiss Kappa statistical analysis. The data is deemed to be statistically significant if the p-value is less than 0.05. In addition, accuracy, precision, recall, and f1 score values will be computed to measure the performance of recognition model.

ELIGIBILITY:
Inclusion Criteria:

* Children aged <18 years old
* Suspected of having hypospadias (hypospadias group)
* Diagnosed as not having hypospadias (control group)

Exclusion Criteria:

* History of hypospadias repair
* Refusal to participate in the study

Max Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The diagnosis of having hypospadias (or not) is established via clinical examination by a pediatric urologist.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-14 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of The Digital Pattern Recognition Model | 1 month
  Accuracy of the digital pattern recognition model compared to clinical assessment by pediatric urologists in measuring:
  1. Hypospadias status: hypospadias or non-hypospadias
  2. Meatal location: glanular, coronal, distal shaft, proximal shaft, penoscrotal
  3. Meatal shape: normal, abnormal
  4. Quality of the urethral plate: good, bad
  5. Glans diameter: in mm
  6. Glans shape: normal, abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Irfan Wahyudi, MD, PhD, Principal Investigator — Department of Urology, Faculty of Medicine, Universitas Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turk E, Guven A, Karaca F, Edirne Y, Karaca I. Using the parents' video camera for the follow-up of children who have undergone hypospadias surgery decreases hospital anxiety of children. J Pediatr Surg. 2013 Nov;48(11):2332-5. doi: 10.1016/j.jpedsurg.2013.04.012. PMID 24210208
- [Background] Han JH, Lee JH, Jun J, Park MU, Lee JS, Park S, Song SH, Kim KS. Validity and reliability of a home-based, guardian-conducted video voiding test for voiding evaluation after hypospadias surgery. Investig Clin Urol. 2020 Jul;61(4):425-431. doi: 10.4111/icu.2020.61.4.425. Epub 2020 Jun 19. PMID 32666000
- [Background] Fernandez N, Lorenzo AJ, Rickard M, Chua M, Pippi-Salle JL, Perez J, Braga LH, Matava C. Digital Pattern Recognition for the Identification and Classification of Hypospadias Using Artificial Intelligence vs Experienced Pediatric Urologist. Urology. 2021 Jan;147:264-269. doi: 10.1016/j.urology.2020.09.019. Epub 2020 Sep 26. PMID 32991907